CLINICAL TRIAL: NCT02334124
Title: CHOICE Trial: Cellulitis at Home Or Inpatient in Children From ED
Brief Title: Comparing the Intravenous Treatment of Skin Infections in Children, Home Versus Hospital
Acronym: CHOICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Principal Investigator, Laila Ibrahim, Dr Laila Ibrahim, MBBChBAO, PhD Student, Murdoch Childrens Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HREC34254F
Record Dates: First submitted 2015-01-04; First posted 2015-01-08 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Cellulitis
MeSH Terms: conditions — Cellulitis | interventions — Home Care Services; Ceftriaxone; Floxacillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home (Experimental): Patients will be treated at home through the Hospital-In-The-Home program with intravenous once daily ceftriaxone (50mg/kg once daily), administered by a nurse/doctor visiting once daily.
  Interventions: Other: Home; Drug: ceftriaxone
- Ward (Active Comparator): Patients will be admitted to hospital ward and treated with six hourly flucloxacillin (50mg/kg), administered by a ward nurse as per routine practice.
  Interventions: Other: Ward; Drug: flucloxacillin

INTERVENTIONS:
Other: Home — The main intervention is for children with uncomplicated cellulitis to remain at home throughout the period of intravenous treatment but as it is not feasible to administer flucloxacillin four times a day by the Hospital-In-The-Home team, once daily ceftriaxone is the most ideal antibiotic to be given to this group
  Arms: Home
Other: Ward — Admission to a hospital based ward
  Arms: Ward
Drug: ceftriaxone — 50mg/kg once daily
  Arms: Home
Drug: flucloxacillin — 50mg/kg 6 hourly
  Arms: Ward

SUMMARY:
Many children every year present to the Emergency Department (ED) at The Royal Children's Hospital (RCH) with cellulitis (skin infection). If it is mild, the children can go home with oral antibiotic treatment. If it is complicated and severe, these children are admitted to hospital for intravenous (IV, through a drip) antibiotic treatment. There is a middle group with uncomplicated moderate/severe cellulitis who require IV antibiotics but who are not acutely unwell. In order to determine whether it is just as effective for children with uncomplicated moderate to severe cellulitis to receive antibiotic treatment at home (via Hospital-In-The-Home) as it is to receive antibiotic treatment in hospital, there is a need to conduct a larger study and randomly assign children to receive either HITH or hospital ward care.

The primary research question to be addressed is:

In children with moderate/severe uncomplicated cellulitis, is the failure rate at 2 days following the first dose of antibiotic non-inferior for children treated with IV antibiotics at home compared to the failure rate at 2 days following the first dose for children treated with IV antibiotics in hospital?

DETAILED DESCRIPTION:
INTRODUCTION AND BACKGROUND Adults with cellulitis commonly have IV antibiotics administered as outpatients, whereas most children are admitted to hospital. Based on a small amount of literature, it is known that some children with moderate/severe cellulitis can also be safely be treated at home.This study will include all children with uncomplicated moderate/severe cellulitis and will therefore demonstrate whether all children with uncomplicated moderate/severe cellulitis can be effectively treated at home.

If the study demonstrates that it is just as effective to treat these children in the home, it has the potential to impact on the child and family's quality of life (QOL) as well as hospital resource management.

PRIMARY OBJECTIVE To compare the failure rate of IV antibiotic treatment of children treated at home (iv ceftriaxone) with those treated in hospital (iv flucloxacillin) in the first 2 days of treatment following the first dose given in the ED in children with moderate/severe cellulitis (Moderate/severe: defined in this study, as those assessed by ED doctor to need iv antibiotics)

SECONDARY OBJECTIVES

To compare:

Time to no progression of cellulitis Time to discharge: number of days (including fractions of days) from the time of arrival in ED to the time the patient no longer needs hospital-based interventions/care, whether in hospital or at home Readmission rate Representation to ED Length of stay in ED Duration of IV antibiotics Rates of IV cannula needing at least one resiting Complications of cellulitis: development of abscess requiring drainage after starting IV antibiotics, bacteraemia Adverse events

Microbiology:

* Rate of ceftriaxone susceptibility in bacteria isolated from a nasal or skin swab of the affected area
* Rate of S. aureus nasal carriage (methicillin-sensitive and methicillin-resistant) collected within 48 hours, after 7-14 days, 3 months and 1 year after starting antibiotics
* Rate of resistant bacteria present in stool samples collected within 48 hours, after 7-14 days, 3 months and 1 year after starting antibiotics. Rates of clinical infection with resistant organisms up to 1 year after starting antibiotics

Differential effect of narrow spectrum (flucloxacillin) and broad spectrum (ceftriaxone) on the nasal and gastrointestinal microbiome from nasal swabs and stool samples collected within 48 hours, after 7-14 days, 3 months and 1 year after starting antibiotics.

Costs of hospital versus HITH treatment: including costs of beds, consumables, nursing and medical time, and overheads including administrative time, information technology, use of hospital cars Quality of life (QOL) indicators Clinical assessments of cellulitis in terms of presence of systemic features, surface area affected (longest length axis multiply by the longest perpendicular axis measured in cm2), severity of swelling (judged by clinician as any one of the following: mild, moderate or severe), intensity of erythema (judged by clinician from a scale of 0 to 5, 0=no erythema and 5=severe and whether the function of the affected area is impaired

STUDY METHODOLOGY ED clinicians (senior doctors, junior doctors or nurse practitioners) will identify patients with moderate/severe cellulitis presenting to RCH ED, at the point of triage or during clinical assessment. The consent will be for randomization, data collection and follow up which is not part of routine practice. Randomisation to the location of treatment is the essential difference from normal clinical practice. Where parents do not give consent, the ED clinician will make the decision on where the patient should be treated.

INTERVENTIONS Although in this proposed study the intervention is treating children at home, currently, based on the prospective observational study, 50% of children with uncomplicated moderate/severe cellulitis are already being sent home by ED clinicians to receive daily IV antibiotics at home. The only new intervention is the randomisation process which will provide a high level of evidence for this practice which has become a standard practice in ED. The researcher or ED clinician will have access to randomization software and perform the randomisation process. Patients who are randomised to HITH will be prescribed iv ceftriaxone (50mg/kg once daily) as per current practice and those randomised to the ward will be prescribed iv flucloxacillin (50mg/kg 6 hourly). On insertion of the IV cannula, the ED clinician will obtain a blood culture. If there is skin breakdown, a skin swab would be done as per routine clinical practice. Prior to commencing IV antibiotics. In addition, the researcher or ED clinician will ask parents to take 2 photos of the cellulitis area using their own camera/phone (if available) after the affected area is demarcated with indelible ink with a tape measure placed along side the area affected. This will be helpful for the reviewing doctor the following day to judge whether there is an improvement.

The first dose of antibiotics will be commenced in ED. For children assigned to hospital ward treatment, the child will be transferred to the ward and the IV infusion continued. Children assigned to the HITH will complete their first dose in ED before going home. The management after this point will be as per usual practice. The responsible ward doctor will review and make all management decisions for patients admitted to the ward whereas the HITH registrar will review the patients on HITH. The research assistant (RA) (a paediatric registrar) will meet with the child and their parent(s) within 24 hours of consent being obtained to answer any further questions parents or participants may have about the study.

Currently, there are no guidelines on when to start IV antibiotic in cellulitis. The investigators' recommendation is provided under section 'Inclusion criteria' and this reflects consensus among RCH ED clinicians. Some patients who did not require IV antibiotics may be recruited but they will exist in both groups.

A nasal swab and stool sample will be requested at four different time points: 1) within 48 hours of the first antibiotic dose; 2) 7-14 days after starting antibiotics; 3) 3 months after starting antibiotics; and 4) 1 year after starting antibiotics. At each time point, additional information will be collected: previous overseas travel, previous hospital admissions, household member who has been admitted to hospital overseas, other antibiotic use, other infections, medical visits or hospital admissions. These samples are optional and do not affect participation in the study.

As per normal practice, patients will be switched to oral therapy after 2-4 days of IV antibiotics, when there is clinical improvement of the cellulitis. Based on the current prospective study, both HITH patients and ward patients are switched to oral antibiotics when there is a reduction in fever, swelling, erythema and improvement of function of affected area (eg. Previously limping, now walking). Once changed to oral antibiotics (as per RCH clinical practice guidelines; cephalexin 25mg/kg 6 hourly, total dose may be combined and divided to twice daily), patients are usually discharged from hospital care and normally not followed up any further in hospital. In this study, the investigators are offering all participants a follow up in clinic 7-14 days (by the RA who is a paediatric registrar) after discharge from hospital. Parents will be requested to bring a stool sample from the patient to the clinic review but this is not mandatory.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 18 years
* Children presenting to RCH ED with moderate/severe cellulitis
* Moderate/severe: defined in this study, as those assessed by ED clinician to need IV antibiotics
* Reasons for starting IV antibiotics include:

  1. Failed oral therapy (not improving despite 24h of oral therapy)
  2. Rapidly spreading redness (from patient/parent history)
  3. Significant swelling/redness/pain
  4. Systemic symptoms/signs (eg. fever, lethargy)
  5. Difficult to treat areas (eg. face, ear, toe)

Exclusion Criteria:

Children will be excluded:

1. With orbital cellulitis or unable to exclude orbital cellulitis,
2. With penetrating injury/bites,
3. With suspected fasciitis or myositis,
4. With toxicity: tachycardia when afebrile or hypotension (both as per the limits set out by RCH Resuscitation Card), poor central perfusion (capillary refill >2 seconds)
5. With immunosuppression,
6. With varicella,
7. With suspected/confirmed foreign body,
8. With abscess not drained,
9. With dental abscess,
10. With concurrent sinusitis or otitis media or lymphadenitis necessitating different antibiotic treatment to flucloxacillin monotherapy or ceftriaxone monotherapy,
11. With liver co-morbidities
12. With other medical diagnoses warranting admission to hospital for observation or treatment relating to the known medical condition
13. With difficult intravenous access,
14. Age <6 months old,
15. Who could be managed on oral antibiotics (ie assessed as mild cellulitis)

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 190 (Actual)
Dates: Start 2015-01; Primary Completion 2017-06 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
Treatment failure (inadequate clinical improvement, adverse event) | Within 2 days of commencing empiric antibiotic
  The primary outcome is failure of treatment defined as no clinical improvement of cellulitis within 2 days of treatment from the start of the first antibiotic dose given in the ED. Any change of initial empiric antibiotics within 2 days from commencement due to:
  * inadequate clinical improvement or
  * adverse events as determined by treating physician will be considered a treatment failure.

SECONDARY OUTCOMES:
Time to no progression | Within 3 days
  Number of days (including fractions of days) elapsed from the start of the first dose in ED (Day 1) to the time at which the cellulitis stops spreading past the marked area, judged during daily assessment of cellulitis
Time to discharge | 14 days
  Number of days (including fractions of days) elapsed from the time of arrival in ED to the moment the patient is discharged.
  (Discharge is defined as when patients admitted to hospital are deemed not to require any hospital funded care/intervention from a hospital based nurse/doctor. The time and date is registered on the electronic hospital database IBA. Admission to hospital is defined as patients who are deemed to need hospital funded care/intervention from a hospital based nurse/doctor)
Readmission rate | 28 days
  Number of children readmitted to hospital within 14 days of discharge date due to the same cellulitis
Representation to ED | 28 days
  Number of children representing to ED within 14 days of discharge and diagnosed to have incomplete resolution or recurrence of same cellulitis
ED Length of stay | 2 days
  Length of stay in ED (from first presentation in ED to time the patient leaves ED to go either home or to ward)
Duration of iv antibiotics | 14 days
  Number of days (including fractions of days) elapsed from the start of the first dose in ED (Day 1) to the time of the last dose
IV cannula resiting (Rates of iv cannula needing at least one resiting) | 14 days
  Rates of iv cannula needing at least one resiting
Complications of cellulitis (Development of abscess requiring drainage) | 14 days
  Development of abscess requiring drainage after starting IV antibiotics and bacteremia
Adverse events | 14 days
  Occurrences of anaphylaxis, allergic reaction (suspected or confirmed) necessitating change of empiric antibiotic, sepsis, death
Comparing patient costs | 14 days
  Comparing ward patient costs and HITH patient costs
Quality of life (QOL) indicators | 1 year
  Quality of life (QOL) indicators (through survey asking parents/patients how much admission to hospital or HITH disrupt their routine)
Cellulitis clinical score | 14 days
  Clinical assessment in all study participants in terms of presence of systemic features, surface area affected (longest length axis multiply by the longest perpendicular axis measured in cm2), severity of swelling (judged by clinician as any one of the following: mild, moderate or severe), intensity of erythema (judged by clinician from a scale of 0 to 5, 0=no erythema and 5=severe erythema), impairment of function of affected area, tenderness of cellulitis area (judged by clinician from a scale of 0 to 5, 0=not tender and 5=very tender).
Microbiology | 1 year
  * Rate of ceftriaxone susceptibility in bacteria isolated from a nasal or skin swab of the affected area
  * Rate of S. aureus nasal carriage (methicillin-sensitive and methicillin-resistant) collected within 48 hours, after 7-14 days, 3 months and 1 year after starting antibiotics
  * Rate of resistant bacteria present in stool samples collected within 48 hours, after 7-14 days, 3 months and 1 year after starting antibiotics. Rates of clinical infection with resistant organisms up to 1 year after starting antibiotics. This outcome may be published separately as require longer follow up.

OTHER OUTCOMES:
Microbiome | 1 year
  • Differential effect of narrow spectrum (flucloxacillin) and broad spectrum (ceftriaxone) on the nasal and gastrointestinal microbiome from nasal swabs and stool samples collected within 48 hours, after 7-14 days, 3 months and 1 year after starting antibiotics. This outcome will be published separately.

CONTACTS AND LOCATIONS:
Overall Officials: Laila F Ibrahim, MBBChBAO, Principal Investigator — Royal Children's Hospital
Locations (1):
- The Royal Children's Hospital Melbourne, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ibrahim LF, Huang L, Hopper SM, Dalziel K, Babl FE, Bryant PA. Intravenous ceftriaxone at home versus intravenous flucloxacillin in hospital for children with cellulitis: a cost-effectiveness analysis. Lancet Infect Dis. 2019 Oct;19(10):1101-1108. doi: 10.1016/S1473-3099(19)30288-9. Epub 2019 Aug 13. PMID 31420292
- [Derived] Ibrahim LF, Hopper SM, Orsini F, Daley AJ, Babl FE, Bryant PA. Efficacy and safety of intravenous ceftriaxone at home versus intravenous flucloxacillin in hospital for children with cellulitis (CHOICE): a single-centre, open-label, randomised, controlled, non-inferiority trial. Lancet Infect Dis. 2019 May;19(5):477-486. doi: 10.1016/S1473-3099(18)30729-1. Epub 2019 Mar 7. PMID 30853250
- [Derived] Ibrahim LF, Babl FE, Orsini F, Hopper SM, Bryant PA. Cellulitis: Home Or Inpatient in Children from the Emergency Department (CHOICE): protocol for a randomised controlled trial. BMJ Open. 2016 Jan 11;6(1):e009606. doi: 10.1136/bmjopen-2015-009606. PMID 26754176